CLINICAL TRIAL: NCT06526949
Title: The Effect of Reiki on Pain, Anxiety and Haemodynamic Parameters in Patients Receiving Mechanical Ventilator Support: A Randomised, Single-Blinded and Placebo-Controlled Study
Brief Title: The Effect of Reiki on Pain, Anxiety and Haemodynamic Parameters in Patients Receiving Mechanical Ventilator Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Yasemin Karacan, Assis.Prof, University of Yalova
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YKaracan
Record Dates: First submitted 2024-07-05; First posted 2024-07-30 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: İntensive Care; Nursing; Reiki
Keywords: Reiki; Critical care; İntensive care; Nursing care
MeSH Terms: interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: Reiki application was performed by a responsible researcher who has a Level 3 (Reiki Master) certificate. To prevent contamination between patients and to provide a suitable environment during the intervention, a curtain-screen system was used in the intensive care unit, and patients were fitted with earplugs to provide a quiet environment during the procedure. During the treatment (total time 30 minutes) the Reiki practitioner gently placed his/her hands on or above the patient's head and eyes, upper body from neck to pelvic area, arms and legs (standard Reiki hand positions).ion time, intensive care unit stay and hemodynamic stability.
  Placebo Control Group In the placebo (sham Reiki) group, treatments were performed by sham practitioners (not involved in the study) who had no experience with energy work and did not believe in energy therapy.
Who Masked: Care Provider
Masking Description: It will not be possible for the researcher to be blinded due to the Reiki application and data collection forms. Blinding in the study will be performed only at the assignment-randomisation stage. Patients will be assigned to the intervention and control groups by the third person (preferably the nurse in charge of intensive care) who is not involved in the research according to the random numbers table in the database sent by the statistician, in the order of group 1 and group 2, using the blinding method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Reiki application was performed by a responsible researcher who has a Level 3 (Reiki Master) certificate. To prevent contamination between patients and to provide a suitable environment during the intervention, a curtain-screen system was used in the intensive care unit, and patients were fitted with earplugs to provide a quiet environment during the procedure. During the treatment (total time 30 minutes) the Reiki practitioner gently placed his/her hands on or above the patient's head and eyes, upper body from neck to pelvic area, arms and legs (standard Reiki hand positions). The application was limited and performed once due to the rapid changes in intubation time, intensive care unit stay and haemodynamic stability.
  Interventions: Behavioral: Reiki
- Placebo Control Group: (Placebo Comparator): In the placebo (sham Reiki) group, treatments were performed by sham practitioners (not involved in the study) who had no experience with energy work and did not believe in energy therapy. To ensure blinding during the sham application, patients received the same hand movements as the experimental group for the same duration. To minimize distractions to the patients during the application, the area was separated by a curtain and screen system, and earplugs were used. The sham practitioner gently placed his hands on or above the patient's head and eyes, upper body from the neck to the pelvic area, arms and legs for 30 minutes. The application was simulated like standard Reiki hand positions.
  Interventions: Other: (Sham Reiki)

INTERVENTIONS:
Behavioral: Reiki — Reiki application was performed by a responsible researcher who has a Level 3 (Reiki Master) certificate. To prevent contamination between patients and to provide a suitable environment during the intervention, a curtain-screen system was used in the intensive care unit, and patients were fitted with earplugs to provide a quiet environment during the procedure. During the treatment (total time 30 minutes) the Reiki practitioner gently placed his/her hands on or above the patient's head and eyes, upper body from neck to pelvic area, arms and legs (standard Reiki hand positions). The application was limited and performed once due to the rapid changes in intubation time, intensive care unit stay and hemodynamic stability.
  Arms: Intervention group
Other: (Sham Reiki) — n the placebo (sham Reiki) group, treatments were performed by sham practitioners (not involved in the study) who had no experience with energy work and did not believe in energy therapy. In order to ensure blinding during the sham application, the patients were given the same hand movements as the experimental group for the same duration. In order not to distract the patients during the application, the area was separated with a curtain and screen system and earplugs were used. The sham practitioner gently placed his hands on or above the patient's head and eyes, upper body from the neck to the pelvic area, arms and legs for 30 minutes. The application was simulated in a manner similar to standard Reiki hand positions.
  Arms: Placebo Control Group:

SUMMARY:
Patients receiving mechanical ventilation (MV) support in intensive care units (ICU) may have some negative experiences. The most common of these are problems such as pain, agitation, anxiety, deterioration in comfort, dry mouth, thirst, and inadequacy in communication.

Reiki, one of the energy therapies among the non-pharmacological nursing practices that have become widespread in recent years, is one of the healing therapies that contribute to the protection and promotion of well-being, healthy aging, and the treatment of some health deviations and is applied noninvasively with hands.

In the literature, there are many studies suggesting that Reiki has positive effects on pain, anxiety and stress response (heart rate, blood pressure, respiratory rate) in patients with Reiki. It is known that these studies generally consist of health professionals such as cancer, haemodialysis, patients undergoing laparoscopic or endoscopic procedures, haemodialysis patients or nurses. Studies have shown that Reiki is especially effective in cancer patients, preoperative stress, anxiety, postoperative pain and symptom management in chronic diseases. For Reiki application in the intensive care unit, only a few studies conducted in the neonatal intensive care unit were found.

DETAILED DESCRIPTION:
The study will consist of 40 patients hospitalized in intensive care units of Yalova Training and Research Hospital and who are receiving mechanical ventilation treatment. The sample will consist of patients who receive mechanical ventilation support in the intensive care unit, who are over 18 years of age, who are willing to participate in the study, who do not have neurological and psychiatric diagnoses, who are not due to drug/alcohol etc. intoxication, who are not in the terminal period, who are not sedated, who have a Glasgow Coma Scale (GCS) score of 9 and above, who are receiving mechanical ventilation support for more than 48 hours, who are hemodynamically stable (not on high dose inotropic support, etc.), and who have a pain score of 3 and above.

Since there was no previous study similar to our research in the literature, the sample size was calculated as 26 patients in the experimental group and 26 patients in the control group with a large effect size d= 0.8, 5% margin of error (α) and statistical power (1-β) = 0.80 as recommended. To increase the power of the study and assume that there may be losses from the sample group, 30 patients were planned to be included in the study, 30 in the experimental group and 30 in the control group.

ELIGIBILITY:
Inclusion Criteria:

1. over 18 years of age,
2. not have a neurological and psychiatric diagnosis,
3. are not due to drug/alcohol etc. intoxication,
4. are not in the terminal period, who are not sedated,
5. have a GCS score of 9 and above, who receive mechanical ventilation support for more than 48 hours,
6. haemodynamically stable (not on high dose inotrope support, etc.),
7. have a pain score of 3 and above.

Exclusion Criteria:

Patients who do not fulfil the inclusion criteria will be excluded.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Change in pain score measured by the Intensive Care Pain Observation Tool (CPOT) in patients receiving mechanical ventilation support | Baseline and immediately after intervention
  Intensive Care Pain Observation Scale (CPOT): This scale was developed to diagnose pain in ICU patients. The scale consists of four subscales expressing behavioural items such as facial expression, body movements, muscle tension and compliance with ventilation for intubated patients or sounds for extubated patients. Three points and above are considered as pain. Each of the sections is evaluated between 0-2 points and The CPOT score ranges from 0-8; higher scores indicate more pain. The scale assesses facial expression, body movements, muscle tension, and compliance with ventilation.

SECONDARY OUTCOMES:
Change in analgesic requirements | During the 30-minute intervention and 30 minutes post-intervention (total 1 hour)
  Analgesic dose or request recorded from ICU records during and up to 1 hour after intervention.
Change in systolic and diastolic blood pressure | Baseline and immediately after intervention
  Blood pressure (mmHg) measured using standard ICU monitors at baseline and immediately post-intervention.
Change in heart rate | Baseline and immediately after intervention
  Heart rate (beats per minute) measured using standard ICU monitors at baseline and immediately post-intervention.
Change in respiratory rate | Baseline and immediately after intervention
  Respiratory rate (breaths per minute) measured using standard ICU monitors at baseline and immediately post-intervention.
Change in anxiety score measured by the Face Anxiety Scale (FAS) | Baseline and immediately after intervention
  Anxiety level was assessed using the Face Anxiety Scale (FAS), which ranges from 1 (no anxiety) to 5 (severe anxiety) based on five standardized facial expressions. The scale has been validated for use in intensive care patients.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Karacan, Principal Investigator — University of Yalova
Locations (1):
- Bursa Training and Research Hospital, Bursa, Yıldırım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The results of the study will be presented after the end of the study.
Supporting Information: Study Protocol, CSR
Time Frame: 07.2025
Access Criteria: The results of the study will be presented after the end of the study.
URL: https://saglikbilimleri.yalova.edu.tr/

REFERENCES:
- [Background] Gokdere Cinar H, Alpar S, Ilhan S. Evaluation of the Impacts of Reiki Touch Therapy on Patients Diagnosed With Fibromyalgia Who Are Followed in the Pain Clinic. Holist Nurs Pract. 2023 May-Jun 01;37(3):161-171. doi: 10.1097/HNP.0000000000000497. Epub 2022 Jan 31. PMID 37070840
- [Derived] Karacan Y, Parlak AG, Ertem AC. Effect of Reiki on Pain, Anxiety, and Hemodynamic Parameters in Mechanically Ventilated Patients: A Randomized, Single-Blind, and Placebo-Controlled Trial. J Integr Complement Med. 2025 Oct 6. doi: 10.1177/27683605251384808. Online ahead of print. PMID 41051913